CLINICAL TRIAL: NCT04403204
Title: Real-time Fluorescence-based Measurement of Bone Perfusion in Post-traumatic Infection
Brief Title: ICG Fluorescence Imaging in Post-traumatic Infection
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other); University of Maryland, Baltimore (Other); University of California, Irvine (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Ida Leah Gitajn, Physician, Dartmouth-Hitchcock Medical Center
Other Study IDs: D20057; 1R01AR077157-01 (NIH)
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Trauma Injury
Keywords: Immunofluorescence; Orthopaedic; Trauma; Infection
MeSH Terms: conditions — Accidental Injuries; Wounds and Injuries; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Established SSI Fracture Cohort: Patients 18 years of age or older. Extremity fracture. Prior definitive fracture management with external fixation, internal fixation, or joint fusion. Superficial, deep, or organ space SSI (as per CDC criteria) at the fracture site that requires operative management. Will have all fracture care surgeries performed by a participating surgeon or delegate. Provision of informed consent
  Interventions: Other: Immunofluorescence Imaging
- Established SSI Fracture Cohort Subset (DCE-MRI): Patients 18 years of age or older. Extremity fracture. Prior definitive fracture management with external fixation, internal fixation, or joint fusion. Superficial, deep, or organ space SSI (as per CDC criteria) at the fracture site that requires operative management. Will have all fracture care surgeries performed by a participating surgeon or delegate. Provision of informed consent
  Interventions: Other: Immunofluorescence Imaging; Other: DCE-MRI

INTERVENTIONS:
Other: Immunofluorescence Imaging — Patients will be administered FDA approved ICG through intravenous injection and imaged by a FDA approved surgical microscope (Spy Elite) which is 0.5 meter away from the subject. Both ICG fluorescence and the two imaging systems have been used for routine clinical practice for many years. Figure (a) shows the Schematic sketch of the imaging systems. ICG fluorescence imaging utilizes intravenously injected ICG, which is a fluorescent dye that is FDA-approved for clinical use, illuminated with near-infrared light. The ICG dye is indirectly activated and the dynamic fluorescence due to bone perfusion can be captured by a video rate imaging system.
Other: DCE-MRI — Characterize the relationship between bone perfusion as quantified by ICG based DCE-FI and DCE-MRI in human patients to develop an accurate depth-sensitive fluorescence imaging model that will correct for the surface-weighted feature of fluorescence imaging
  Groups: Established SSI Fracture Cohort Subset (DCE-MRI)

SUMMARY:
The focus of this prospective observational study is to (1) establish the range and variation associated with bone/soft tissue perfusion in fracture patients, using ICG fluorescence imaging; (2) examine the relationship between perfusion and complications such as surgical site infection (SSI), persistent SSI, and fracture nonunion; (3) to determine whether the quantitative ICG fluorescence can be used to guide bony debridement in the setting of infected fracture to minimize complications.

DETAILED DESCRIPTION:
This will be a prospective observational trial to better understand the range and variation associated with bone/soft tissue perfusion in fracture patients and examine the relationship between perfusion, measured using quantitative Indocyanine green (ICG) fluorescence and complications such as surgical site infection (SSI), persistent SSI, and fracture nonunion. Primary outcome measure is complication (either infection, recurrent infection or nonunion).

Eligible consenting patients will receive standard of care treatment for their fracture or infection including irrigation and debridement of their operative site and/or fracture fixation. After exposure, 0.1 mg/Kg ICG will be injected intravenously and video rate ICG fluorescence images will be acquired 20 seconds before and 4 minutes after the injection, each before and after debridement.

A subset of 30 post-fracture complication patients will undergo surgical treatment for their infection in Center of Innovation Surgery (CIS) and have either an intraoperative Dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) after exposure but before the ICG injection or a preoperative DCE-MRI. Patients receiving surgery in the CIS will be required to sign an additional CIS-specific consent document.

The need for repeat surgical procedure will be left up to the treating surgeon. If repeat procedure is needed, pre- and post-debridement quantitative ICG fluorescence images will be obtained at each procedure.

Study participants will be followed at 2 weeks, 6 weeks, 3 months, 6 months, and one year from their index study surgery. Complication including index infection, recurrent infection or delaying union/nonunion will be identified at the time of diagnosis and/or during each participants assessment that occurs during routine outpatient clinic visit. Detailed information on the infection including date of diagnosis, participant signs and symptoms, culture test results, method of treatment(s), and date of resolution will be documented.

ELIGIBILITY:
Inclusion Criteria:

Established SSI Fracture (Cohort Cohort 1, Group 1)

1. Patients 18 years of age or older.
2. Extremity fracture.
3. Prior definitive fracture management with external fixation, internal fixation, or joint fusion.
4. Superficial, deep, or organ space SSI (as per CDC criteria) at the fracture site that requires operative management.
5. Will have all fracture care surgeries performed by a participating surgeon or delegate.
6. Provision of informed consent.

Subset: DCE-MRI (Cohort 1-1, Group 2)

1. Patients 18 years of age or older.
2. Closed extremity fracture.
3. Planned definitive fracture management with external fixation, internal fixation, or joint fusion.
4. Will have all planned fracture care surgeries performed by a participating surgeon or delegate.
5. Provision of informed consent.

Exclusion Criteria:

Established SSI Fracture Cohort (Cohort 1, Group 1)

1. Fracture of the hand.
2. Iodine allergy.
3. Received previous surgical debridement to manage the SSI.
4. Incarceration.
5. Problems, in the judgment of study personnel, with maintaining follow-up with the patient.

   Subset: DCE-MRI (Cohort 1-1, Group2)
6. the presence of an electronic implant, such as a pacemaker
7. the presence of a metal implant, such as an aneurysm clip
8. the presence of other contraindication(s), as determined by the MRI technologists and radiologists.
9. A history of allergy to iodides
10. A GFR < 30 ml/min as determined by blood test on the day of NIR/MR imaging, or from lab results within 3 months of DCE-MRI for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older who present with SSI following fracture or joint fusion Established SSI fracture cohort (Cohort 1). A subset of Cohort 1 will be considered for the Subset DCE-MRI cohort (Cohort 1-1).
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing post procedure surgical site infections | 1 year
  Post-procedure surgical site infection using CDC criteria will be documented at each follow-up appointment up to one year
Number of patients requiring unplanned fracture-related reoperations | 1 year
  All unplanned reoperations will be documented

CONTACTS AND LOCATIONS:
Overall Officials: Ida L Gitajn, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (4):
- United States (4):
  - University of California, Irvine, Irvine, California
  - University of Maryland, Baltimore R. Adams Cowley Shock Trauma, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire

IPD SHARING:
Plan to Share IPD: No